CLINICAL TRIAL: NCT04529915
Title: Multicenter Clinical Research for Early Diagnosis of Lung Cancer Using Blood Plasma
Brief Title: Multicenter Clinical Research for Early Diagnosis of Lung Cancer Using Blood Plasma Derived Exosome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hyun Koo Kim, Professor, Korea University Guro Hospital
Other Study IDs: 2020GR0176
Record Dates: First submitted 2020-08-02; First posted 2020-08-28 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Lung Cancer
Keywords: Blood plasma; Exosome; Liquid biopsy; Lung cancer; Biomarker; Deep-learning analysis
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer
  Interventions: Diagnostic Test: Exosome sampling
- Healthy
  Interventions: Diagnostic Test: Exosome sampling

INTERVENTIONS:
Diagnostic Test: Exosome sampling — * Centrifugation of blood plasma
  * Size exclusion chromatography
  * ELISA assay, Western blotting
  * Deep-learning analysis

SUMMARY:
Lung cancer is a leading cause of cancer death worldwide. Early diagnosis is linked to a better prognosis. Further, surgical resection at the early stages of non-small cell lung cancer (NSCLC) results in markedly improved survival rates. Computed tomography (CT)- or bronchoscopy-guided needle biopsies are standard definitive diagnostic procedures for lung cancer and are used to obtain tissue for pathological examination. However, these procedures are invasive, difficult to repeat, expensive, and risk exposure to radiation. Conversely, liquid biopsies, such as circulating tumor cells (CTCs), circulating tumor DNA (ctDNA), and extracellular vesicles (EVs), are simple and less invasive procedures that can be repeated more frequently than tissue biopsies.

To analyze the exosomes abundantly present in the blood and to conduct clinical studies to determine whether it is possible to diagnose lung cancer. To this end, blood samples from normal people (n = 150) and lung cancer patients (n = 320) are obtained from the Human biobank of five hospitals participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary adenocarcinoma of lung with permanent pathology of N0 or N1
2. Patients with T1mi, Tsi, T1a, T1b, T1c, T2a, and T2b stage
3. An adult of Korean nationality
4. Patients without prior chemo/radiation treatment prior to lung cancer surgery
5. Patients who have not been diagnosed with other cancers prior to lung cancer surgery

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this study, Koreans, regardless of gender, were studied for adults over 40 years of age.
  Participating institutions for this clinical research are Korea University Guro Hospital, Gangnam Severance Hospital, Bundang Seoul National University Hospital, Seoul Asan Hospital, and Samsung Seoul Hospital.
  Blood plasma samples is taken from stored in the biobank of each hospital.
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the distinction between healthy controls and lung cancer patients through deep-learning analysis of exosomes | 3 years
  Comparative evaluation of whether it is possible to distinguish between healthy controls and lung cancer patients through deep-learning analysis of exosomes
Evaluating the possibility of distinguishing between normal and lung cancer patients through the analysis of lung cancer-specific exosomal protein | 3 years
  Quantitative analysis using lung cancer-specific exosomal protein evaluated the possibility of distinguishing between healthy controls and lung cancer patients.

SECONDARY OUTCOMES:
Evaluation of the possibility of distinguishing the early pathological stages in lung cancer patients through deep-learning analysis of exosomes | 3 years
  Evaluating whether the early stages of lung cancer patients can be distinguished using deep-learning analysis of exosomes
Evaluation of the possibility of distinguishing the early pathological stages in lung cancer patients through quantitative analysis of lung cancer specific exosomal proteins | 3 years
  Evaluating whether the early stages of lung cancer patients can be distinguished using quantitative analysis of lung cancer specific exosomal proteins

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Koo MD, PhD, MD, PhD, Principal Investigator — Professor
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaplan RN, Rafii S, Lyden D. Preparing the "soil": the premetastatic niche. Cancer Res. 2006 Dec 1;66(23):11089-93. doi: 10.1158/0008-5472.CAN-06-2407. PMID 17145848
- [Background] Psaila B, Lyden D. The metastatic niche: adapting the foreign soil. Nat Rev Cancer. 2009 Apr;9(4):285-93. doi: 10.1038/nrc2621. PMID 19308068
- [Background] Talmadge JE, Fidler IJ. AACR centennial series: the biology of cancer metastasis: historical perspective. Cancer Res. 2010 Jul 15;70(14):5649-69. doi: 10.1158/0008-5472.CAN-10-1040. Epub 2010 Jul 7. PMID 20610625
- [Background] Bidard FC, Pierga JY, Vincent-Salomon A, Poupon MF. A "class action" against the microenvironment: do cancer cells cooperate in metastasis? Cancer Metastasis Rev. 2008 Mar;27(1):5-10. doi: 10.1007/s10555-007-9103-x. PMID 18066649
- [Background] van Akkooi AC, Verhoef C, Eggermont AM. Importance of tumor load in the sentinel node in melanoma: clinical dilemmas. Nat Rev Clin Oncol. 2010 Aug;7(8):446-54. doi: 10.1038/nrclinonc.2010.100. Epub 2010 Jun 22. PMID 20567244